CLINICAL TRIAL: NCT03596619
Title: The Study of Plum-blossom Needling Enhancing Efficacy of Aminolevulinic Acid-photodynamic Therapy for Actinic Keratosis: a Randomized and Multi-center Clinical Trial
Brief Title: The Study of Plum-blossom Needling Enhancing Efficacy of Aminolevulinic Acid-photodynamic Therapy for Actinic Keratosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Dermatology Hospital (Other)
Collaborators: Peking University People's Hospital (Other); Xiangya Hospital of Central South University (Other); Central South University (Other); Wuhan No.1 Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Tripler Army Medical Center (U.S. Federal Agency); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Chinese PLA General Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Xiuli Wang, Institute of Photomedicine, Shanghai Dermatology Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-05
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Actinic Keratoses
Keywords: plum-blossom needling; Photodynamic Therapy; Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBN-ALA-PDT Group (Experimental): The PBN-ALA-PDT group underwent vertical skin tapping with PBN before applying 10% ALA cream and narrow-band light-emitting diode (LED) irradiation (mean 633 nm, with a standard deviation [SD] of 10 nm; 100-200 J/cm2).
  Interventions: Device: PBN
- ALA-PDT Group (No Intervention): The ALA-PDT group received ALA cream and irradiation only.

INTERVENTIONS:
Device: PBN — The PBN-ALA-PDT group underwent vertical skin tapping with PBN before applying 10% ALA cream and narrow-band light-emitting diode (LED) irradiation (mean 633 nm, with a standard deviation [SD] of 10 nm; 100-200 J/cm2). The ALA-PDT group received ALA cream and irradiation only.
  Arms: PBN-ALA-PDT Group

SUMMARY:
Background Limited in the depth of absorption and penetration of photosensitizers, ALA-PDT treatment is not strong enough for thickening significantly AK lesions. Pre-study has proved that plum-blossom needling facilitates delivery of topical ALA into the dermis. It could help ALA to diffuse a little more broadly in superficial dermis and obtain similar clinical effect with a much lower cost.

Objective We sought to investigate whether plum-blossom needling (PBN) would enhance the efficacy of ALA-PDT for AKs.

Methods Two hundred and fifty patients, previously diagnosed as having AKs of the face and scalp, were randomized distribution into two groups. The PBN-ALA-PDT group underwent vertical skin tapping with PBN before applying 10% ALA cream and narrow-band light-emitting diode (LED) irradiation (mean 633 nm, with a standard deviation [SD] of 10 nm; 100-200 J/cm2). The ALA-PDT group received ALA cream and irradiation only. During the next 1 year period of follow up, patients were clinically evaluated for new AKs.

ELIGIBILITY:
Inclusion Criteria:

* (1) Clinical diagnosed with AK (OLSEN classification grade I, II, III), aged > 18 years (Because no dosing or adverse event data are currently available on the use of topical aminolevulinic acid in patients <18 years of age, children are excluded from this study); (2) All patients are unfit and reluctant to undergo surgery for any reasons, and volunteered to participate in the study and ability to understand and the willingness to sign a written informed consent. Patents are willing to pay for the treatment, and agreed to take a picture of the skin lesions.

Exclusion Criteria:

* (1) Those who had ALA-PDT and any other studies that affect this study within 12 weeks ; (2) There are other facial diseases that may affect the efficacy evaluation, such as other photodermatosis; (3) Take phototoxic or photosensitizer within 8 weeks; (4) clinical and / or pathological prove that the tumor has invaded other organs or tissues; (5) Serious immunocompromised persons; (6) scar constitution; (7) Patients are known to have skin photosensitivity, porphyria, or allergies to ALA, light or lidocaine; (8) Persons are suffering from severe internal diseases, mental and mental illness, infectious diseases or pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The clearance rate of Actinic Keratoses | two weeks after first session
  The change rate in lesion clearance of Actinic Keratoses at two weeks after the first session will be measured as the primary outcome

SECONDARY OUTCOMES:
Treatment sessions | two weeks after the last session
  Number of treatment sessions required for clinical cure
Number of new Actinic Keratoses | 1, 3, 12 months after last session
  The change in number of actinic keratoses at each follow-up will be measured as the second outcome
Adverse events | 1, 3, 12 months after last session
  Measurement of crusting, erythema, edema, pain and et al.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Wang, PhD, MD, Study Chair — Shanghai Skin Disease Hospital
Locations (2):
- China (2):
  - Shanghai Dermatology Hospital, Shanghai, Jingan
  - Xiuli Wang, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
underlie results
Supporting Information: CSR
Time Frame: One year after finishing this study and for permanency
Access Criteria: anyone who search pubmed
URL: http://www.ncbi.nlm.nih.gov/pubmed

REFERENCES:
- [Result] Pomerantz H, Hogan D, Eilers D, Swetter SM, Chen SC, Jacob SE, Warshaw EM, Stricklin G, Dellavalle RP, Sidhu-Malik N, Konnikov N, Werth VP, Keri J, Lew R, Weinstock MA; Veterans Affairs Keratinocyte Carcinoma Chemoprevention (VAKCC) Trial Group. Long-term Efficacy of Topical Fluorouracil Cream, 5%, for Treating Actinic Keratosis: A Randomized Clinical Trial. JAMA Dermatol. 2015 Sep;151(9):952-60. doi: 10.1001/jamadermatol.2015.0502. PMID 25950503
- [Result] Chen J, Zhang Y, Wang P, Wang B, Zhang G, Wang X. Plum-blossom needling promoted PpIX fluorescence intensity from 5-aminolevulinic acid in porcine skin model and patients with actnic keratosis. Photodiagnosis Photodyn Ther. 2016 Sep;15:182-90. doi: 10.1016/j.pdpdt.2016.06.012. Epub 2016 Jun 30. PMID 27375183
- [Result] Jia XH, Liu LN. [Plum blossom needling for 74 cases of scapulohumeral periarthritis]. Zhongguo Zhen Jiu. 2011 Nov;31(11):1040. No abstract available. Chinese. PMID 22136038
- [Result] Yao ZH, Yao XL, Wan SQ. Observation on 52 cases of paralysis of common peroneal nerve treated by acupuncture and plum-blossom needling. J Tradit Chin Med. 1984 Jun;4(2):97-100. No abstract available. PMID 6567734